CLINICAL TRIAL: NCT06460662
Title: Effects of Agility and Perturbation Based Training in Addition to Routine Physical Therapy on Pain, Function and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Effects of Agility and Perturbation Based Training in Addition to Routine Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0193 Maryam
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: pain; function; quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agility and perturbation training group (Experimental): Group A will receive agility and perturbation training techniques in addition to the same routine physical therapy as Group B.
  The Agility training exercises include:
  * Side Stepping
  * Braiding Activities
  * Front and Back Crossover Steps During Forward Ambulation
  * Multiple Changes in Direction During Walking on Therapist Command
  The perturbation training exercises include:
  * Double-Leg Foam Balance Activity
  * Tilt board Balance Training
  * Rollerboard and Platform Perturbations
  Interventions: Other: Routine Physical Therapy
- Routine physical therapy (Active Comparator): Group B: Routine physical therapy Group that includes:
  * Calf Stretching
  * Hamstring Stretching
  * Prone Quadriceps Stretching
  * Long-Sitting Knee Flexion and Extension
  * Quadriceps setting
  * Supine Straight Leg Raises
  * Prone Hip Extensions
  * Standing Hamstring Curls With Cuff Weights
  * Standing Calf Raises
  * Treadmill Walking
  * Mobilization techniques
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Routine Physical Therapy — Group B: Routine physical therapy Group that includes:
  * Calf Stretching
  * Hamstring Stretching
  * Prone Quadriceps Stretching
  * Long-Sitting Knee Flexion and Extension
  * Quadriceps setting
  * Supine Straight Leg Raises
  * Prone Hip Extensions
  * Standing Hamstring Curls With Cuff Weights
  * Standing Calf Raises
  * Treadmill Walking
  * Mobilization techniques

SUMMARY:
Osteoarthritis is a degenerative joint disease. Knee OA patients sometimes report episodes of knee instability that limit their ADLs. The episodes of instability are similar to those reported in knee ligament injuries. It is believed that modifications of interventions that are used to promote knee stability in knee ligament injuries can be used in knee OA to enhance knee stability and function. The purpose of this study will be to determine the effects of agility and perturbation-based training in addition to routine physical therapy on pain, function, quality of life and disability in knee osteoarthritis.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Al Syed Touqeer Altaf Surgical Hospital through a convenience sampling technique on 26 patients, which will be allocated using computer-generated randomization into two groups. Group A will be treated with agility and perturbation training techniques in addition to the same routine physical therapy as Group B, and Group B will receive only routine physical therapy. Outcome measures will be conducted through NPRS, WOMAC, SF-36, and KOS-ADLs questionnaires. All the outcome measures will be assessed pre and post-treatment, and the assessor will be blind. Frequency of the treatment will be 3 sessions per week for 4 weeks. Data will be analyzed using SPSS software version 25.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female.
* Subjects with Kellgren and Lawrence grade II and III osteoarthritis.
* OA diagnosed subjects according to American College of Rheumatology ACR criteria;

  * Morning stiffness ≤ 30 minutes.
  * Crepitus with active motion of the knee (while weight bearing).
  * Tenderness to palpation of the bony margins of the joint, bony enlargement, and no palpable warmth.

Exclusion Criteria:

* Ligament or meniscal injury around the knee.
* Suffering from acute synovitis
* Neuromuscular disorders.
* Cognitive impairments.
* Required use of an assistive device for ambulation.
* Reported a history of 2 or more falls within the previous year.
* Undergone total knee arthroplasty.
* Uncontrolled hypertension, history of cardiovascular disease, neurological disorders that affected lower extremity function.
* Severe visual problems.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Numeric pain rate scale (NPRS) | upto 4 weeks
  Numeric pain rate scale will be used to quantify patient level of pain. The Numeric Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The common format is a horizontal bar or line. Although various iterations exist, the most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from (no pain at all) to 10 (worst imaginable pain) i.e. higher scores indicating greater pain intensity. High test-retest reliability has been observed in both literate and illiterate patients with rheumatoid arthritis (r = 0.96 and 0.95, respectively) before and after medical consultation. For construct validity, the NPRS was shown to be highly correlated with the VAS in patients with rheumatic and other chronic pain conditions (pain>6 months): correlations range from 0.86 to 0.95.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | upto 4 weeks
  Patients' knee function and stiffness will be measured through the Western Ontario and McMaster Universities Arthritis Index (WOMAC) . It is a self-administered questionnaire consisting of 24 items divided into 3 subscales; Pain-5 items, Stiffness-2 items, Physical Function-17 items .
  WOMAC Index was developed in 1982 at Western Ontario and McMaster Universities. WOMAC is available in over 65 languages and has been linguistically validated. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually, a sum of the scores for all three subscales gives a total WOMAC score.
SF-36 (Short form) | upto 4 weeks
  36-Item Short Form Survey (SF-36) will be used to assess the quality of life. (SF-36) is an outcome measure instrument that is often used, a well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study, which is an objective measure of quality of life. It comprises 36 questions that cover eight domains of health. The 36 questions on the SF-36 are meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health.Possible scores range from 0 to 100, with higher scores representing better health status.
Knee Outcome Survey Activities of Daily Living KOS-ADLS | upto 4 weeks
  Knee outcome survey ADLS will be used to measure disability. The ADLS is a 14 item scale that queries patients about how their knee symptoms effect their ability to perform general daily activities (6 items) as well as how their knee condition effects their ability to perform specific functional tasks (8 items). Each item is scored 0-5 with 5 indicating "no difficulty" and 0 representing "unable to perform". The highest possible score is 70. The scores of all items are summed, divided by 70, and then multiplied by 100 to give an overall ADLS percent rating. Higher percentages reflect higher levels of functional ability.
  The ADLS demonstrated high test-retest reliability in 52 subjects with knee pathology. The ICC score for test-retest reliability over a 24 hour period was .97. Construct validity was determined through correlations with the Lysholm Knee Scale (r = .78 to .86).

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Ijaz, MSPT*, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Sher Shah Road, Shadbagh, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lange AK, Vanwanseele B, Fiatarone Singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Rheum. 2008 Oct 15;59(10):1488-94. doi: 10.1002/art.24118. PMID 18821647
- [Background] Hicks-Little CA, Peindl RD, Hubbard-Turner TJ, Cordova ML. The Relationship Between Early-Stage Knee Osteoarthritis and Lower-Extremity Alignment, Joint Laxity, and Subjective Scores of Pain, Stiffness, and Function. J Sport Rehabil. 2016 Aug;25(3):213-8. doi: 10.1123/jsr.2014-0170. Epub 2016 Jul 21. PMID 27445119
- [Background] Michael JW, Schluter-Brust KU, Eysel P. The epidemiology, etiology, diagnosis, and treatment of osteoarthritis of the knee. Dtsch Arztebl Int. 2010 Mar;107(9):152-62. doi: 10.3238/arztebl.2010.0152. Epub 2010 Mar 5. PMID 20305774
- [Background] Samson DJ, Grant MD, Ratko TA, Bonnell CJ, Ziegler KM, Aronson N. Treatment of primary and secondary osteoarthritis of the knee. Evid Rep Technol Assess (Full Rep). 2007 Sep;(157):1-157. PMID 18088162
- [Background] Collins NJ, Hart HF, Mills KAG. Osteoarthritis year in review 2018: rehabilitation and outcomes. Osteoarthritis Cartilage. 2019 Mar;27(3):378-391. doi: 10.1016/j.joca.2018.11.010. Epub 2018 Dec 7. PMID 30529739
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Jamtvedt G, Dahm KT, Christie A, Moe RH, Haavardsholm E, Holm I, Hagen KB. Physical therapy interventions for patients with osteoarthritis of the knee: an overview of systematic reviews. Phys Ther. 2008 Jan;88(1):123-36. doi: 10.2522/ptj.20070043. Epub 2007 Nov 6. PMID 17986496
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766